CLINICAL TRIAL: NCT05367141
Title: Active (CDSS) Control Blinded Multicenter, Cluster-randomized Trial of the Adherence to Clinical Practice Guidelines Using the Clinical Decision Support System in Patients With Hypertension and Atrial Fibrillation (INTELLECT II Trial)
Brief Title: Improvement Adherence to Clinical Practice Guidelines Using the Clinical Decision Support System in Patients With Hypertension and Atrial Fibrillation
Acronym: INTELLECTII
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samara Regional Cardiology Dispensary (Other)
Collaborators: Medicbook LLC (Unknown)
Responsible Party: Principal Investigator, Prof. Dmitry Duplyakov FESC, Ass. Prof. Dmitry Duplyakov M.D.,Ph.D., Samara Regional Cardiology Dispensary
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SamaraRCD
Record Dates: First submitted 2022-01-11; First posted 2022-05-10 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Atrial Fibrillation; Arterial Hypertension
Keywords: clinical practice guidelines; Clinical Decision Support Systems; adherence to guidelines; evidence-based medicine
MeSH Terms: conditions — Atrial Fibrillation; Hypertension

STUDY DESIGN:
Intervention Model Description: multicenter, cluster-randomized, single-blind, controlled study with blinded outcome assessment.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CDSS (Active Comparator): patient management with aid of CDSS
  Interventions: Other: CDSS ("MedicBK")
- standart care (No Intervention): patient management with standard care according to guidelines

INTERVENTIONS:
Other: CDSS ("MedicBK") — Clinical decision support system ("MedicBK") is a computer-based program that analyzes published evidence and provides prompts and reminders to assist health care providers in implementing clinical guidelines and science-based medicine at the point of care.
  Arms: CDSS

SUMMARY:
The Clinical Decision Support Systems (CDSS) based on real clinical data and its own algorithms can help to make the right choice according to guidelines. The goal of the INTELLECT II study is to investigate treatment adherence to guidelines/science-based medicine and its impact on patient outcomes into two groups of doctors, clinical centers with standard care of treatment (control), and clinical centers using CDSS (active).

DETAILED DESCRIPTION:
Hypertension and atrial fibrillation are 2 important public health priorities. There is a gap between evidence-based best management and actual clinical practice. To decrease this gap, clinical practice guidelines (CPGs), based on available evidence are employed. Clinical decision support system ("MedicBK") is a computer-based program that analyzes published evidence and provides prompts and reminders to assist health care providers in implementing clinical guidelines and science-based medicine at the point of care. The INTELLECT II trial is designed as a multicenter, cluster-randomized, single-blind, controlled study with blinded outcome assessment. Approximately 10 centers from Russia will be enrolled. Centers managing patients with symptomatic atrial fibrillation and/or hypertension will be randomized to either patient management with aid of CDSS ("MedicBK") or standard care.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years old
* Patients diagnosed with nonvalvular atrial fibrillation and hypertension and indications for therapy according to European guidelines.

Exclusion Criteria:

* Inability to adhere to study procedures
* Severe heart-valve disorder
* Stroke within 14 days or severe stroke within 6 months before screening
* Active bleedings
* Thyroid dysfunction
* Pregnancy
* Secondary hypertension

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 282 (Actual)
Dates: Start 2022-05-17 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2023-08-22 (Actual)

PRIMARY OUTCOMES:
Compliance with AF/hypertension clinical practice guidelines | 1 month
  number of patients treated in accordance with current ESC clinical guidelines for management atrial fibrillation evaluated by independent professionals compared with Clinical decision support system MedicBK

SECONDARY OUTCOMES:
Total cardiovascular events | 6 months
  total stroke or systemic embolism, total coronary heart disease, major bleeding, recurrence of atrial fibrillation, hospitalization or death from congestive heart failure and other significant vascular deaths
Total mortality | 6 months
  death from all causes
total number of non-planing visits and hospitalization | 6 months
  non-planing hospitalizations, non-planning visits, urgent visits

CONTACTS AND LOCATIONS:
Locations (1):
- Samara Regional Cardiology Dispansery, Samara, Russia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Duplyakov D.V., Shebonkina D.A., Uranov A.E., Mikheenko I.L., Astrakova K.S., Gartung A.A., Adonina E.V., Tukhbatova A.A., Kuzmin V.P., Fedorova G.A., Gabidullova D.A., Skuratova M.A., Shechovtsova T.A., Losik D.V. Optimizing compliance with clinical guidelines using a clinical decision support system in patients with hypertension and atrial fibrillation in real-world practice: a cluster-randomized comparative study INTELLECT-2. Russian Journal of Cardiology. 2025;30(12):6365. (In Russ.) https://doi.org/10.15829/1560-4071-2025-6365. EDN: OKIRDC
- See also: Related Info — https://doi.org/10.15829/1560-4071-2025-6365